CLINICAL TRIAL: NCT05980819
Title: Workshops in Sustainable Healthcare: Assessing the Utility of Expert-led Teaching in Aiding the Clinical Implementation of Sustainable Quality Improvement Principles
Brief Title: Workshops in Sustainable Healthcare to Assess How Teaching Can Aid Core Principle Implementation
Acronym: WISH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LHS0018
Record Dates: First submitted 2023-02-08; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-01

CONDITIONS: Quality Improvement; Medical Education
Keywords: Sustainability; Medical Education; Healthcare

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Volunteers (Experimental): All volunteers will partake in this educational study at the same timepoints, there will be no blinding, but there will be an unbiased recruitment effort
  Interventions: Other: Sustainability lecture and opportunity to create a project

INTERVENTIONS:
Other: Sustainability lecture and opportunity to create a project — Pure education

SUMMARY:
With more frequent extreme weather events, climbing atmospheric Carbon dioxide and unabated use of fossil fuels, planetary health and sustainability will become crucial to future medical practice. Clinical educators must rise to the challenge, educating and empowering tutees to ensure their understanding of green healthcare principles and solutions.

Research at the University College London and the Universities of Bristol and Exeter has been conducted into engaging medical students with the theory of sustainability. What has not been explored is how to have them engage with the topic practically, providing them with frameworks and opportunities to their knowledge into practical scenarios. What we propose is a short study conducted over the period of a month in October 2023 that pairs educational sessions to answer the research question: do practical workshops help to cement sustainable teaching for attendees, help them bring out their individual ideas and experience surrounding sustainability, and empower them to implement comparable solutions in their clinical practice? Historically, these projects have ignored multidisciplinary practice. Specialists of any grade in any field can practice sustainability. As such, any healthcare student/professional is eligible, pending their consent. To facilitate this broad eligibility base, and to bring diversity of ideas to the workshops, both students at Liverpool University and any interested staff at the Liverpool University Hospitals Foundation Trust will be eligible for the project.

Following a pre-session questionnaire to gauge baseline, participants will be taught the core principles of clinical sustainability in a remote 2-hour, interactive lecture-based session. This would be followed up by a hybrid 2-hour practical workshop session later that week. Here, those consenting to attend will have a chance to work through different clinical scenarios with experts in different fields. Each session will have feedback forms to gauge compounding of knowledge, engagement and empowerment, our primary outcome measures.

DETAILED DESCRIPTION:
A research participant will be either a health professional of any denomination based at the Liverpool University Hospitals Foundation Trust (LUHFT) or a medical/allied healthcare student based at the University of Liverpool, Liverpool John Moores or Edge Hill.

They will be granted access to an online consent form through formal distribution through the Trust/Medical School and through posters placed around the Trust. This will inform them about the project's intentions and what may happen to their data during the course of the project, thus allowing them to opt-in to the project as needed.

The study design itself is that of a cohort study with subsequent quantitative and qualitative analysis of various descriptive features of the participant cohort. Specifically, we will assess participant baselines - their rates of exposure to sustainability principles in healthcare between their different specialties, their knowledge of quality improvement methodology and experience in its application - in addition to their confidence in the understanding of sustainability principles in healthcare, as well as their confidence in their ability to apply it to clinical scenarios. This is in line with the 4-point Kirkpatrick model for training evaluation, covering reaction, learning, behaviour and results.

Our null hypothesis is that there will be no significant difference in confidence applying sustainable healthcare principles in clinical practice after the workshop based teaching versus before, as well as no significant difference in rates of exposure between specialties or knowledge of quality improvement methodology.

The study itself will be conducted over a two-session period in late September through to early October across 18/09/23 to 16/10/23, lasting ideally no longer than three to four weeks (pending site availability for study rooms). It will be split into an education session conducted in a hybrid manner, whereby QI methodology and its relationship to sustainability is taught through didactic lectures to a combined in person and online audience. Participants will then be encouraged to create their own sustainable QI project plan using this methodology, and then would attend an expert-led set of workshops (hybrid, online and in person) where breakout groups from the initial cohort are assigned experts (volunteers from or beyond the Trust with expertise in sustainable healthcare, attending in person or online depending on availability) to have their work critiqued formally and to discuss implementation techniques for the idea in clinical practice. Using pre-determined mark schemes created by the PI, the team will also receive input from the trainers themselves to ascertain student engagement with the teaching, the viability of their created projects and extent to which they successfully implemented the core taught principles in their project designs.

This will be preceded by a month's worth of recruitment from 07/08/23 ending on 04/09/23 by which potential participants will be able to access the aforementioned consent form either online through formally provided links or the posters, thus being able to opt-in to the project. Researcher bias will be avoided through unbiased recruitment, not conducted directly by the researchers but by intermediaries so as to not choose individuals that may already have experience, for example. Participants will be given the choice as to whether to opt in the research. There is no limit on the upper sample size of the cohort, though for the purposes of efficient and worthwhile breakout rooms for the experts, a minimum sample of 20 would be required (approximately 10 students and 10 healthcare professionals employed by LUHFT). This should be sufficient for the descriptive analyses required from a statistical perspective.

Statistical analysis will be conducted in a mixed manner assessing frequencies, associations and qualitative themes. Cronbach's alpha will be used to assess internal consistency and reliability of the pre and post session questionnaires. Differences between students' pre- and post-session scores will be analysed using chi-squared tests. Qualitative data will be coded into themes relating to outcomes, processes, and suggestions for improvement, facilitated by NVivo13 software. Statistical theory has been discussed with a senior statistician prior to its inclusion on these forms.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare students at the University of Liverpool/Liverpool John Moores/ Edge Hill who are assigned placement at the LUHFT Trust:

  * medical students
  * nursing students
  * dental students
  * student paramedics
  * student occupational therapists
  * student physiotherapists
  * student radiographers
  * student dieticians
  * operating department practitioners
  * student speech and language therapists
  * student psychologists
  * student pharmacists
* NHS Doctors
* Junior doctors from FY1 to ST8, including SAS doctors or Doctors not in Training
* Senior Clinical Fellows
* Consultant Doctors
* NHS Healthcare professionals of any description

  * Nurses (any band)
  * Dentists (any grade)
  * Psychologists (any band)
  * Pharmacists (any band)
  * Paramedics (any grade)
  * Occupational Therapists (any band)
  * Physiotherapists (any band)
  * Radiographers (any band)
  * Dieticians (any band)
  * Operating department practitioners (any band)
  * Speech and language therapists (any band)

Exclusion Criteria:

* Those who are not healthcare students from the institutions above
* Those who are not NHS Healthcare Staff members from the LUHFT Trust

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Confidence in applying sustainable healthcare principles to clinical scenarios following the lectures and expert-led workshop. | 4 weeks. To be assessed during the pre-course survey in the month prior to the first session, then to be assessed after the second session (the post-course survey will cover both sessions and will be available for a month, being delivered to participants
  Confidence level as measured on a Likert Scale of 1-5 with 1 being unconfident, and 5 being highly confident. Comparison will be made using a pre-session Likert scale and a post-session Likert scale addressing the same question. Statistically, non-parametric tests such as Mann-Whitney U will be used to generate results.

SECONDARY OUTCOMES:
Presence of difference in baseline knowledge of sustainability principles between different healthcare professional types and students in the region | 4 weeks. To be assessed during the pre-course survey in the month prior to the first session, then to be assessed after the second session (the post-course survey will cover both sessions and will be available for a month, being delivered to participants
  Knowledge level as measured on a Likert Scale of 1-5 with 1 being Very poor, and 5 being exceptional. Comparison will be made using a pre-session Likert scale and a post-session Likert scale addressing the same question. However, this in particular is a categorical binary variable - yes/no - as we want to see if there is a difference or not, which is different to the extent of difference.
Presence of difference in confidence in applying sustainability principles in practice between different healthcare professional types and students in the region | 4 weeks. To be assessed during the pre-course survey in the month prior to the first session, then to be assessed after the second session (the post-course survey will cover both sessions and will be available for a month, being delivered to participants
  Confidence level as measured on a Likert Scale of 1-5 with 1 being unconfident, and 5 being highly confident. Comparison will be made using a pre-session Likert scale and a post-session Likert scale addressing the same question. However, this in particular is a categorical binary variable - yes/no - as we want to see if there is a difference or not, which is different to the extent of difference.
Extent of difference in improvement in knowledge of core sustainability principles between different groups (students versus professionals) | 4 weeks. To be assessed during the pre-course survey in the month prior to the first session, then to be assessed after the second session (the post-course survey will cover both sessions and will be available for a month, being delivered to participants
  Knowledge levels as measured on a Likert Scale of 1-5 with 1 being Very poor, and 5 being exceptional for each feature. Comparative outcome measure between different groups - Wilcoxon signed-rank and Mann-Whitney U tests to be used to generate comparative results between different groups and the same group (unpaired and paired).
Extent of difference in improvement in confidence in applying sustainable principles in practice between different groups (students versus professionals) | 4 weeks. To be assessed during the pre-course survey in the month prior to the first session, then to be assessed after the second session (the post-course survey will cover both sessions and will be available for a month, being delivered to participants
  Confidence levels as measured on a Likert Scale of 1-5 with 1 being unconfident, and 5 being highly confident for each feature. Comparative outcome measure between different groups - Wilcoxon signed-rank and Mann-Whitney U tests to be used to generate comparative results between different groups and the same group (unpaired and paired).
Assessing a single taught session's value in guiding a participant's ability to create a clinically viable project using objective criteria as devised by the PI | 4 weeks. Markers to complete their assessments prior to the second session - they would then feed back individually to participants during the sessions. They can take up to a month to deliver the emails to the participants via their collected emails.
  Comparative outcome measure between individuals regardless of background Assessing a single taught session's value in guiding a participant's ability to create a clinically viable project using objective criteria
  Comparative outcome measure between individuals regardless of background Mark scheme has been created by the PI. It covers likely success of the project submitted across 4 key criteria (health impact, environmental impact, social impact and feasibility) across a 6-point Likert scale (negligible impact being the most negative outcome for a given criterion, followed by minor impact, average impact, above average impact, exceptional impact and not applicable). Consideration of the Core Features of Clinical Sustainability, as presented to participants within the teaching itself, will be assessed using the same key criteria and scaling. Qualitative feedback will also be collected from the markers under 'any other comments' and themed based on overarching results.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Jukka, MBChB, Study Chair — Royal Liverpool University Hospital
Locations (1):
- Royal Liverpool University Hospital, Liverpool, Merseyside, United Kingdom